CLINICAL TRIAL: NCT07070596
Title: NATURCEL Registry: Study of the NATURal History, Epidemiological, Clinical, Diagnostic and Therapeutic Aspects of CELiac Disease and Non-celiac Enteropathies
Brief Title: Study of the NATURal History, Epidemiological, Clinical, Diagnostic and Therapeutic Aspects of CELiac Disease and Non-celiac Enteropathies
Acronym: NATURCEL
Status: Recruiting | Type: Observational
Sponsor: Hospital Mutua de Terrassa (Other)
Collaborators: Centro de Investigación Biomédica en Red de enfermedades hepáticas y digestivas (CIBERehd) (Unknown); Hospital Universitari de Bellvitge (Other); Hospital Clinic of Barcelona (Other); Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina (Other); Hospital Arnau de Vilanova (Other)
Responsible Party: Sponsor
Other Study IDs: P/25-076
Record Dates: First submitted 2025-06-12; First posted 2025-07-17 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-06

CONDITIONS: Celiac Disease
Keywords: Gluten-Related Disorders; Gluten-Free Diet; HLA-DQ2; HLA-DQ8; Tissue Transglutaminase Antibodies; Anti-Endomysial Antibodies; Pediatric and Adult Celiac Disease; TCRγδ+ lymphocytes
MeSH Terms: conditions — Celiac Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with suspected celiac disease

SUMMARY:
Celiac disease is a chronic immune-mediated enteropathy triggered by gluten intake, which affects the small intestine in genetically susceptible subjects (HLA-DQ2 and/or HLA-DQ8). Affecting both children and adults, it is among the most common genetically determined disorders in Western countries. The disease is characterized by clinical manifestations (mainly digestive symptoms and signs of intestinal malabsorption), the presence of specific antibodies (tissue transglutaminase and endomysium) and enteropathy. Currently, the only treatment for celiac disease is a strict gluten-free diet for life.

The main objective of the NATURCEL registry (Study of the NATURal history, epidemiological, clinical, diagnostic and therapeutic aspects of celiac disease and non-celiac enteropathies) is to collect a wide range of data (epidemiological, clinical, genetic, immunological, etc.) for scientific and translational purposes.

The registry will include individuals diagnosed with celiac disease or other gluten-related disorders, as well as patients with non-celiac enteropathies evaluated for suspected celiac disease. In the future, the project also aims to establish a biobank-an organized repository of biological samples-to further support scientific and medical research in this field.

ELIGIBILITY:
Inclusion Criteria:

* Individuals under diagnostic evaluation for celiac disease

Exclusion Criteria:

* Failure to sign informed consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Individuals diagnosed with celiac disease and other gluten-related disorders based on established diagnostic guidelines (2019 European Society for the Study of CD for Adults, the Paris Consensus Criteria for the Diagnosis of Seronegative CD, and the 2020 ESPGHAN Criteria for the Diagnosis of CD in Childhood) and individuals with non-celiac enteropathies who have been found in the diagnostic process of suspected celiac disease.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2030-01-01 (Estimated); Study Completion 2030-01-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with confirmed celiac disease diagnosis based on serologic and histologic criteria among those with suspected celiac disease | End of diagnostic evaluation (up to 10 weeks after inclusion)

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitari MútuaTerrassa, Terrassa, Barcelona, Spain